CLINICAL TRIAL: NCT06418880
Title: Automated Insulin Delivery for Inpatients With Dysglycemia (AIDING) Randomized Controlled Trial
Brief Title: Automated Insulin Delivery for Inpatients With Dysglycemia
Acronym: AIDING
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Francisco Pasquel, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007081; 1R01DK138366-01 (NIH); 2025P012163 (Other: Emory IRB)
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: continuous glucose monitoring; automated insulin delivery; Insulin Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (Active Comparator): The control group will follow the hospital's usual practice for subcutaneous insulin for glucose control. It will be managed by the admitting team with the assistance of an inpatient endocrine team.
  Participants will wear a real-time CGM for 10 days or until hospital discharge (if <10 days)
  Interventions: Combination Product: Standard of Care Insulin Therapy + CGM
- Intervention (Experimental): Participants in the intervention arm will be assigned to the Omnipod 5 AID system with integrated Dexcom CGM. These devices will communicate with a patient-specific smartphone secured within the patient room and remotely monitored by the nursing station.
  Nursing staff on medical-surgical units will provide insulin therapy using the investigational device for participants randomized to the intervention arm, including delivering insulin boluses, monitoring CGM values and trends, validating CGM accuracy against POC glucose, and performing routine device exchanges (Pod or CGM) when indicated AID therapy will continue for 10 days or until hospital discharge (if <10 days)
  Interventions: Device: AID system with Remote Real-Time CGM

INTERVENTIONS:
Device: AID system with Remote Real-Time CGM — The Omnipod 5 AID System is comprised of two components:
  * Omnipod 5 Pod (insulin infusion pump with SmartAdjust technology)
  * Omnipod 5 App (installed on the Controller or smart phone) The Omnipod 5 AID pod is a lightweight, self-adhesive device that the user fills with U-100 rapid-acting insulin and wears directly on their body. The Pod delivers insulin into the user's body through a small flexible tube, called a cannula, based on the commands from the compatible Controller. In the Omnipod 5 AID System, the Pod itself houses the MPC algorithm and communicates directly with the CGM and the Omnipod 5 App. Based on predicted glucose values, the algorithm commands the Pod's insulin delivery through micro-boluses.
  Arms: Intervention
Combination Product: Standard of Care Insulin Therapy + CGM — This includes the usage of subcutaneous insulin for glucose control. Participants will wear a real-time Continuous Monitoring (CGM) for 10 days or until hospital discharge (if <10 days).
  Treatment decisions will be based on POC testing with consideration of daily evaluation of CGM patterns.
  Other Names: Multiple Daily Injections +CGM
  Arms: Control

SUMMARY:
This randomized controlled trial will test the efficacy and safety of automated insulin delivery (AID) in hospitalized patients with diabetes (type 1 or type 2) requiring insulin therapy who are admitted to general medical/surgical floors.

The main objectives of this study are:

* To test the efficacy and safety of AID versus multiple daily insulin injections (MDI) + CGM in the inpatient setting
* To determine differences in CGM-derived metrics between AID and MDI plus CGM in the hospital and explore differences in treatment effect according to individual characteristics.

Participants will be:

* Randomized to AID + remote CGM (intervention) or multiple daily insulin injections (MDI) + CGM (control group)
* Followed for a total of 10 days or until hospital discharge (if less than 10 days).

DETAILED DESCRIPTION:
Annually, over 8 million people in the United States are hospitalized due to diabetes. Among these patients, those with uncontrolled diabetes are at a significantly heightened risk for poor hospital outcomes. However, achieving glycemic targets within hospital settings proves challenging, as doing so often increases the risk of iatrogenic hypoglycemia. This is exacerbated by the variable insulin therapy requirements that arise during acute illnesses, such as unpredictable nutrition intake, illness severity, and the effects of various medications. These fluctuations pose a substantial challenge for healthcare providers tasked with caring for patients with diabetes.

The usage of diabetes technology may offer an opportunity to improve inpatient diabetes care, but best practices are not yet defined. The COVID-19 pandemic has highlighted how accelerated use of technologies (e.g., telemedicine, e-consults, and remote monitoring) helps healthcare systems adapt care delivery while minimizing exposure risk. Following the non-objection by the US Food and Drug Administration (FDA) to the use of CGM in the hospital, the investigators and others implemented the usage of remote real-time CGM to treat patients with COVID-19. Initial clinical trials using remote real-time CGM have shown modest improvements in hypoglycemia detection and prevention and minimal or no increases in time spent in the target range (TIR) in non-ICU patients.

The use of AID with remote insulin delivery and remote glucose monitoring is novel for the inpatient setting. The use of AID allows for 288 automated insulin dosing alterations per day, which is infeasible for hospital staff and could help proactively compensate for the multitude of factors affecting insulin requirements in the hospital. Preliminary data from AID trials with a single European AID system (using an insulin pump with tubing) have shown improvements in glycemic control in diverse populations without increasing the risk of hypoglycemia. However, these trials have limited involvement of patient care teams and the feasibility of hospital implementation and adoption is unknown.

Using single-use insulin patch-pumps (without tubing) may offer a unique opportunity for hospital use of AID; however, no randomized controlled data on the use of AID in the hospital is available in the US. Results from our recently completed pilot study show that using AID with remote CGM is feasible in the hospital and appears to be associated with good glycemic control.

In addition to improving glycemic control, this approach will:

* Offer a unique treatment option for patients typically excluded from inpatient clinical trials, including patients with type 1 diabetes, steroids, medical nutrition therapy, or those under isolation precautions.
* Use superficial wearable medical devices to alleviate inconveniences and discomforts to patients associated with current standard-of-care insulin therapy. The combination of a CGM and a patch-based insulin pump can greatly reduce the need for recurrent "sticks" and "pricks." They may thereby improve the quality of experience for patients admitted to the hospital.
* Introduce remote insulin delivery and remote glucose monitoring, offering an unprecedented opportunity for effective diabetes care for people with highly contagious diseases or while interacting with patients during emergency conditions.
* Set the stage for subsequent inpatient diabetes technology implementation efforts. The investigator's approach has multiple layers of safety to ensure improved glycemic control without increasing the risk of hypoglycemia, including a) nursing staff training for rapid response, b) EHR documentation and validation of sensor glucose values to confirm accuracy, c) remote monitoring with alarms (telemetry and inpatient treatment team).

ELIGIBILITY:
Inclusion Criteria:

• Any person ≥18 years of age with diabetes mellitus (except cystic fibrosis- and pregnancy-related) admitted to general (non-ICU) medical-surgical hospital services which require inpatient insulin therapy (i.e.,TID or T2D with ≥2 glucose values ≥180mg/dl)

Exclusion Criteria:

* Patients admitted to ICU
* Patients anticipated to require less than 48 hours admission.
* Current evidence of hyperglycemic crises (diabetic ketoacidosis or hyperosmolar hyperglycemic state)
* Severe anemia with hemoglobin <7 g/dL
* Evidence of hemodynamic instability
* Hypoxia (SpO2 <92% on supplemental oxygen)
* Pre-admission or inpatient total-daily insulin dose >150 units daily
* T2D patients on sliding scale insulin therapy alone (no scheduled basal or bolus insulin) and with glucose levels below 180 mg/dl
* Patients without diabetes with stress hyperglycemia (not related to steroids or medical nutrition therapy) and with HbA1c <6.5%
* Patients on AID as outpatient
* Patients who previously participated in AIDING feasibility trial or this RCT
* Patients with a condition impeding their ability to consent or answer questionnaires or notify staff of symptoms.
* Patients who are pregnant time of enrollment
* Patients who are unable or unwilling to use rapid-acting insulin analogs (Humalog, Admelog, or Novolog) during the study
* Use of hydroxyurea, high dose of acetaminophen (>4 grams/day), or high dose ascorbic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Efficacy: Time spent in glucose target range | Up to 10 days (or hospital discharge if before 10 days)
  This will be captured by the percentage of time spent in glucose target range (TIR 70-180 mg/dl);
Safety: Time spent below the target glucose range | Up to 10 days (or hospital discharge if before 10 days)
  This will be captured by the percentage of time spent below glucose range (TBR <54 mg/dl).

SECONDARY OUTCOMES:
TAR >250mg/dl | Up to 10 days (or hospital discharge if before 10 days)
  Percentage of time spent above 250 mg/dl
TBR <70 mg/dl | Up to 10 days (or hospital discharge if before 10 days)
  Percentage of time spent below range (TBR <70 mg/dl)
Mean hospitalization glucose | Up to 10 days (or hospital discharge if before 10 days)
  This will be calculated as the mean of total glucose levels during the hospital stay.

OTHER OUTCOMES:
Time spent above 180 mg/dl | Up to 10 days (or hospital discharge if before 10 days)
  Percentage of time spent above the glucose levels of 180 mg/dl
Time spent between 70-99 mg/dl | Up to 10 days (or hospital discharge if before 10 days)
  Percentage of time spent between the range of 70-99 mg/dl
Glycemic events above 300 mg/dl | Up to 10 days (or hospital discharge if before 10 days)
  Number of Glycemic events above 300 mg/dl will be captured
Glycemic events below 54 mg/dl | Up to 10 days (or hospital discharge if before 10 days)
  Number of Glycemic events below 54 mg/dl will be captured
Number of hypoglycemic episodes (Glucose <40 mg/dl) | Up to 10 days (or hospital discharge if before 10 days)
  defined as an event that required assistance of another person due to altered consciousness to actively administer parenteral carbohydrate, glucagon, or other resuscitative actions. This means that the participant was impaired cognitively to the point that the participant was unable to drink or eat oral carbs (e.g. juice, crackers), was incoherent, disoriented, and/or combative, or experienced seizure or coma.
Number of Diabetes-related Ketoacidosis Events | Up to 10 days (or hospital discharge if before 10 days)
  The number of Diabetes-related ketoacidosis (DKA) events across all participants.
Number of hyperosmolar hyperglycemic syndrome (HHS) events | Up to 10 days (or hospital discharge if before 10 days)
  The number of hyperosmolar hyperglycemic syndrome (HHS) events across all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Pasquel, M.D., M.P.H, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - Grady Health System (non-CRN), Atlanta, Georgia
  - University of Virginia School of Medicine, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2025-11-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT06418880/SAP_000.pdf
  • Informed Consent Form (2025-10-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT06418880/ICF_001.pdf